CLINICAL TRIAL: NCT01824459
Title: A Randomized, Open, Multi-center, Phase III Study of S-1+Oxaliplatin vs.S-1+Cisplatin First-line Treatment in Advanced or Recurrent Non-intestinal Type Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma Patients
Brief Title: S-1+Oxaliplatin vs.S-1+Cisplatin First-line Treatment of Advanced or Recurrent Non-intestinal Type Gastric Adenocarcinoma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ruihua Xu, vice president of SunYat-sen University Cancer Center,head of medical oncology department, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOX-DGCA
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Gastric Cancer
Keywords: Non-intestinal type gastric cancer; Advance Gastric Cancer; Recurrent Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; SOX, S-1+Oxaliplatin; OS,; ORR,; PFS,; TTF,; safety
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Oxaliplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-1 + cisplatin(SP) (Active Comparator): S-1：40~60mg bid，d1~14 q3W cisplatin：60mg/m2，iv drip ，d1,q3W Number of Cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: S-1; Drug: Cisplatin
- S-1+Oxaliplatin（SOX） (Experimental): S-1：40~60mg bid，d1~14 q3W oxaliplatin：130mg/m2，iv drip for 2h，d1,q3W Number of Cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: S-1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: S-1 — S-1：40~60mg bid，d1~14 q3W
Drug: Oxaliplatin — oxaliplatin：130mg/m2，iv drip for 2h，d1,q3W
  Arms: S-1+Oxaliplatin（SOX）
Drug: Cisplatin — cisplatin：60mg/m2，iv drip ，d1,q3W
  Arms: S-1 + cisplatin(SP)

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of S-1+Oxaliplatin vs.S-1+Cisplatin First-line Treatment in Advanced or Recurrent Non-intestinal Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma Patients.

DETAILED DESCRIPTION:
The primary endpoint is Overall survival time (OS).Secondary endpoints are overall response rate (ORR), time to treatment failure (TTF),progression free survival (PFS)and the adverse reactions(AE) of the two groups .

Study design:

This is a prospective randomized control study.

Sample size:

Sample size considerations were based on the survival end point. The improvement in median survival from 10 months in the S-1+cisplatin arm to 13 months in the S-1+oxaliplatin arm was considered clinically relevant in this patient population. A total of 576 patients were required for a two-tailed log-rank test at the 5% significance and at least 80% power. The planned enrolled time was 48 months and 1 year of follow up, and a drop-out rate of 5%.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed unresectable advanced or recurrent diffuse-type or mixed-type gastric adenocarcinoma or gastroesophageal junction adenocarcinoma.
2. 18 years old to 75 years old, able to conduct oral administration.
3. Measurable disease or non-measurable but evaluable disease, according to the Response Evaluation Criteria in Solid Tumours(RECIST 1.1)
4. No palliative chemotherapy and radiotherapy. Previous adjuvant or neoadjuvant chemotherapy , if applicable, more than 12 months.
5. ECOG systemic status score of 0 to 2.
6. normal organ function, that meet the following criteria:

   1. ALT and AST(≤2.5 times ULN (≤5 times ULN in patients with liver metastases)
   2. ALP ≤ 2 times ULN ; (for patients with liver metastases can be no limit to the ALP).
   3. Total bilirubin ≤ 1 times ULN.
   4. Absolute neutrophil count ≥ 2.0 × 10^9 / L.
   5. Platelet count ≥ 100 × 10^9 / L.
   6. Hemoglobin ≥ 80g / L.
   7. Creatinine ≤ 1.25 times ULN.
   8. The estimated creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula).
7. Signed informed consent, treatment, follow-up and inspection in accordance with the study protocol.
8. Life expectancy greater than 3 months.
9. At least 3 weeks after major surgery.

Exclusion Criteria:

1. Previous adjuvant or neoadjuvant chemotherapy within the prescribed time
2. the investigator determines that the patient is not suitable for participation in this study, and specifically includes (but is not limited to):

   1. The past five years there have been other malignancies, but after appropriate treatment of cervical carcinoma in situ and non-melanoma skin cancer.
   2. brain metastases or leptomeningeal metastasis.
   3. myocardial infarction (within the past six months), severe unstable angina, congestive heart failure.
   4. Serious complications (including paralytic ileus, intestinal obstruction, interstitial pneumonia, lung fibrosis, beyond the control of diabetes, renal insufficiency and cirrhosis of the liver, etc.).
   5. Chronic nausea, vomiting, or diarrhea (per day greater than or equal to 4 times or watery stools).
   6. Gastrointestinal bleeding, and need for frequent blood transfusions.
   7. human immunodeficiency virus (HIV) carrier or suffering from AIDS (AIDS).
   8. Suffering from a mental illness.
   9. neuropathy severity ≥grade 2 .
   10. Infectious disease or inflammation, body temperature ≥ 38 ℃.
3. Cisplatin, oxaliplatin, or S-1 allergy.
4. Pregnancy or breast-feeding women.
5. refused to take appropriate contraceptive measures (including male patients).
6. Under experimental drug within 4 weeks.
7. Under other anti-cancer treatment.
8. HER2 IHC(3+) or IHC(2+) /FISH(+)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2013-04; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1-1.5 year
  OS means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 12 weeks till death or lost

SECONDARY OUTCOMES:
Objective response rate | 1 year
  The primary endpoint is objective response rate,which equals CR+PR.
time to treatment failure (TTF) | 6 months
  The duration is from the randomized time to treatment termination due to any reason. The reasons may include disease progression, treatment toxicity, patient selection or death.
progression-free survival (PFS) | 6 months
  The duration is from the randomized time to disease progression or death due to any reason.
Adverse events (AE) | 1-1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: ruihua xu, Professor, Principal Investigator — SunYat-sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China